CLINICAL TRIAL: NCT03422094
Title: A Pilot Study to Assess the Safety, Feasibility, and Immunogenicity of a Neoantigen-based Personalized Vaccine Combined With Immune Checkpoint Blockade Therapy in Patients With Newly Diagnosed, Unmethylated Glioblastoma
Brief Title: Neoantigen-based Personalized Vaccine Combined With Immune Checkpoint Blockade Therapy in Patients With Newly Diagnosed, Unmethylated Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Manufacturer changed focus to cell therapy
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201804195
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — poly ICLC; Nivolumab; Ipilimumab; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A: NeoVax+Nivolumab (start at time of progression) (Experimental): * NeoVax given on Days 1, 8, 15, and 22 of Cycle 1 (priming phase), and then on Day 1 of each subsequent cycle (boosting phase)
  * Nivolumab 480 mg i.v. given on Day 1 of each cycle beginning at time of progression
  Interventions: Biological: NeoVax; Biological: Nivolumab; Procedure: Research blood draw; Procedure: Leukapheresis for research
- Cohort B: NeoVax+Nivolumab (start with Cycle 2) (Experimental): * NeoVax given on Days 1, 8, 15, and 22 of Cycle 1 (priming phase), and then on Day 1 of each subsequent cycle (boosting phase)
  * Nivolumab 480 mg i.v. given on Day 1 of each cycle beginning with Cycle 2 (start of boosting phase)
  Interventions: Biological: NeoVax; Biological: Nivolumab; Procedure: Research blood draw; Procedure: Leukapheresis for research
- Cohort C: NeoVax + Nivolumab (start with Cycle 1) (Experimental): * NeoVax given on Days 1, 8, 15, and 22 of Cycle 1 (priming phase), and then on Day 1 of each subsequent cycle (boosting phase)
  * Nivolumab 480 mg i.v. given on Day 1 of Cycle 1 (priming phase), and then on Day 1 of each subsequent cycle (boosting phase)
  Interventions: Biological: NeoVax; Biological: Nivolumab; Procedure: Research blood draw; Procedure: Leukapheresis for research
- Cohort D: NeoVax+Ipilimumab+Nivolumab (start with Cycle 3) (Experimental): * NeoVax given on Days 1, 8, 15, and 22 of Cycle 1 (priming phase), and then on Day 1 of each subsequent cycle (boosting phase)
  * Ipilimumab 1 mg/kg i.v. given on Days 1 and 22 of Cycle 1 (priming phase)
  * Nivolumab 480 mg i.v. given on Day 1 of Cycle 3 and then on Day 1 of each subsequent cycle
  Interventions: Biological: NeoVax; Biological: Nivolumab; Biological: Ipilimumab; Procedure: Research blood draw; Procedure: Leukapheresis for research
- Cohort E: NeoVax+Ipilimumab+Nivolumab (day 1&15 each cycle) (Experimental): * NeoVax given on Days 1, 8, 15, and 22 of Cycle 1 (priming phase), and then on Day 1 of each subsequent cycle (boosting phase)
  * Ipilimumab 1 mg/kg i.v. given every 6 weeks beginning on Day 1 of Cycle 1 (C1D1, C2D15, C4D1, C5D15, C7D1, C8D15 …)
  * Nivolumab 3 mg/kg i.v. given on Days 1 and 15 of each cycle (q2w) beginning on Day 1 of Cycle 1
  Interventions: Biological: NeoVax; Biological: Nivolumab; Biological: Ipilimumab; Procedure: Research blood draw; Procedure: Leukapheresis for research

INTERVENTIONS:
Biological: NeoVax — At each vaccination time point, patients will receive up to 20 synthetic long peptides co-administered with 1.5 mg of poly-ICLC divided into a maximum of four injections (pools). Each pool (of vaccine + poly IC:LC) will be administered to one of the four limbs (right axilla, left axilla, right inguina, left inguina) by subcutaneous injection.
  Other Names: Synthetic long peptides plus poly-ICLC
Biological: Nivolumab — Nivolumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: Opdivo
Biological: Ipilimumab — Ipilimumab is a recombinant, human monoclonal antibody that binds to the cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4)
  Other Names: Yervoy
  Arms: Cohort D: NeoVax+Ipilimumab+Nivolumab (start with Cycle 3); Cohort E: NeoVax+Ipilimumab+Nivolumab (day 1&15 each cycle)
Procedure: Research blood draw — -Baseline, cycle 2 day 1, cycle 4 day 1, and time of progression or discontinuation of treatment
Procedure: Leukapheresis for research — -Baseline, cycle 4 day 1, and time of progression or discontinuation of treatment

SUMMARY:
This is a single institution, open-label, multi-arm, pilot study assessing the safety, feasibility, and immunogenicity of a personalized neoantigen-based vaccine plus poly-ICLC (NeoVax) combined with immune checkpoint inhibitors in subjects with newly diagnosed, unmethylated glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically confirmed unmethylated glioblastoma multiforme (WHO grade IV). Patients with secondary glioblastoma, in particular those who are IDH1 or IDH2 mutant, will not be excluded. Unmethylated MGMT must be confirmed by a PCR-based assay.
* Patients who had craniotomy with biopsy, subtotal resection, total gross resection, or re-resection will be permitted.
* Consented to genome sequencing and dbGaP-based data sharing and has provided or will provide germline (PBMC) and tumor DNA/RNA samples of adequate quality for sequencing. (Acquisition of specimens for sequencing and the sequencing itself may be done as part of routine care or another research project.)
* At least 18 years of age.
* Karnofsky performance status ≥ 60%
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Systemic corticosteroid therapy is permitted provided dosing is no greater than 4 mg per day (dexamethasone or equivalent) on the day of vaccine administration.
* Bevacizumab will be allowed if given for symptomatic control of vasogenic edema and to avoid high dose of corticosteroids.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation, including at least 5 months (for women of childbearing potential) and at least 7 months (for men) after last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* As this study aims to assess the immunogenicity of various vaccine plus adjuvant combinations, no prior immunotherapy will be permitted.
* Inadequate tissue acquisition to allow for neoantigen screening.
* No candidate neoantigen identified during screening.
* A history of other malignancy ≤ 3 years previous with the exception of non-melanoma skin cancer, any in situ cancer that has been successfully resected and cured, treated superficial bladder cancer, or any early-stage solid tumor that was successfully resected without need for adjuvant radiation or chemotherapy.
* Receiving any other investigational agents within 4 weeks of beginning study treatment.
* Known allergy, or history of serious adverse reaction to, vaccines such as anaphylaxis, hives, or respiratory difficulty.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to poly-ICLC or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of pre-existing immunodeficiency disorder or autoimmune condition requiring immunosuppressive therapy. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines.
* Presence of clinically significant increased intracranial pressure (e.g. impending herniation) or hemorrhage, uncontrolled seizures, or requirement for immediate palliative treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of first dose of vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-04-26 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of regimen as measured by a <= 33% dose-limiting toxicity (DLT) rate for a given cohort | Up to 90 days after start of treatment
  * The DLT observation period is 60 days after C1D1 for patients enrolled to Cohorts A, C, and D and is 90 days after C1D1 for patients enrolled to Cohorts B and E.
  * DLT is defined as any grade 3 or greater event that occurs during the DLT observation period that is considered at least possibly related to the study treatment.
Feasibility of generating a personalized neoantigen peptide vaccine as measured by the ability to identify candidate tumor-specific neoantigens | From time of resection to 4 weeks post-radiation therapy (approximately 14 weeks)
Feasibility of generating a personalized neoantigen peptide vaccine as measured by the the ability to manufacture a neoantigen-based synthetic long peptide vaccine | From time of resection to 4 weeks post-radiation therapy (approximately 14 weeks)
Feasibility of generating a personalized neoantigen peptide vaccine as measured by the ability to administer the vaccine to a patient at 4 weeks post-completion of radiotherapy | From time of resection to 4 weeks post-radiation therapy (approximately 14 weeks)

SECONDARY OUTCOMES:
Immunogenicity of a personalized neoantigen peptide vaccine as measured by the ability to generate a measurable neoantigen-specific T cell response in vaccinated patients | Week 4 post-vaccination
Immunogenicity of a personalized neoantigen peptide vaccine as measured by the ability to generate a measurable neoantigen-specific T cell response in vaccinated patients | Week 16 post-vaccination
Immunogenicity of a personalized neoantigen peptide vaccine as measured by the number of individual neoantigens per number of neoantigens vaccinated against, with which a measurable T cell-specific response | Week 4 post-vaccination
Immunogenicity of a personalized neoantigen peptide vaccine as measured by the number of individual neoantigens per number of neoantigens vaccinated against, with which a measurable T cell-specific response | Week 16 post-vaccination
Number of high quality candidate neoantigens present in patients with newly diagnosed glioblastoma | Up to 2 weeks post sequencing
  High quality neoantigens will be defined as those that meet criteria for inclusion in a vaccine
Progression-free (PFS) survival rate | 6 months
Overall survival (OS) rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tanner Johanns, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

DOCUMENTS (1):
  • Informed Consent Form (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03422094/ICF_000.pdf